CLINICAL TRIAL: NCT05122728
Title: Post-Concussion Neuromuscular Function and Musculoskeletal Injury Risk
Brief Title: Post-Concussion Musculoskeletal Injury Risks
Status: Recruiting | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Womack Army Medical Center (U.S. Federal Agency); University of Georgia (Other)
Responsible Party: Principal Investigator, Bradford Hendershot, Facility Research Director, Walter Reed National Military Medical Center
Other Study IDs: WRNMMC-2021-0362
Record Dates: First submitted 2021-10-28; First posted 2021-11-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Injury
Keywords: musculoskeletal injury; biomechanics; movement assessment; neuromuscular control; traumatic brain injury; TBI; concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussed Cohort: Active duty Service Members and physically active civilians who have self-reported as asymptomatic post-concussion.
  Interventions: Other: Post-Concussion Neuromuscular Function and Musculoskeletal Injury Risk Assessment
- Non-Concussed Cohort: Gender, age, occupation, and physical activity matched active duty Service Members and physically active civilians who have not sustained a concussion.
  Interventions: Other: Post-Concussion Neuromuscular Function and Musculoskeletal Injury Risk Assessment

INTERVENTIONS:
Other: Post-Concussion Neuromuscular Function and Musculoskeletal Injury Risk Assessment — Participants will complete a comprehensive biomechanical and neuromuscular assessments to elucidate the underlying neuromuscular control mechanisms that may contribute to increased MSKI risk following concussion. Participants will also complete a battery of self-report psychosocial measures.
  Biomechanical Dynamic Movement Assessments:
  * Jump-Landing
  * Single Leg Hop
  * Anticipated Cut
  * Gait - Single Task
  * Gait - Dual Task
  Strength and Voluntary Muscle Activation Assessments:
  * Interpolated Twitch Technique
  * Muscular Ramp Contraction
  Sensory assessments:
  * Proprioception - Closed Chain
  * Passive Joint Repositioning
  * Light Touch Sensation
  Patient Reported Outcomes:
  * Self-Reported Musculoskeletal Injuries
  * National Institutes of Health Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function
  * PROMIS Pain Interference
  * PROMIS Depression
  * PROMIS Anxiety
  * Brief Resilience Scale (BRS)
  * Tampa Scale of Kinesiophobia (TSK-11)

SUMMARY:
Musculoskeletal injuries (MSKI) and traumatic brain injury (TBI) are the signature injuries of the ongoing military conflicts. MSKI affect 800,000 Service Members annually and TBI have impacted more than 350,000 in the past 19 years and account for 22% of all combat casualties. Concussion, a mild form of TBI, increases MSKI risk in physically active individuals, including Service Members.

The overall goal of the study is to identify the neuromuscular control mechanisms that increase MSKI risk following concussion. It is hypothesized that concussed individuals will display abnormal neuromuscular function that increases MSKI risk, as compared to non-concussed controls. The study will employ a multi-center, prospective, case-matched control observational study to identify the differences in neuromuscular function following concussion that may contribute to increased MSKI risk. Once the neuromuscular control mechanisms that increase MSKI risk following concussion are identified, targeted risk mitigation strategies can be developed to reduce MSKI risk.

DETAILED DESCRIPTION:
Musculoskeletal injuries are the greatest unsolved public health problem facing the military and significantly diminish Service member's medical readiness. MSKI affect 800,000 Service members and result in 25 million limited-duty days annually. Additionally, among civilians peers, sport-related MSKI affect as many as 12 million people annually. In total, MSKI place a significant burden on military and civilian populations, with a combined financial burden of more than $980 billion per year in the US alone.

Traumatic brain injuries (TBI), specifically concussions a mild form of TBI, have been classified by the National Institutes of Health and Centers for Disease Control as a "serious health problem" in the US. TBIs have impacted more than 350,000 Service members in the past 19 years. Concussions negatively affect individuals' quality of life, as assessed by patient report outcome (PRO) psychosocial measures, including worse scores for measures of anxiety, depression, fatigue, anger, and pain immediately following concussion, as compared to when they are cleared to return-to-duty/activity (RTD/A).

Musculoskeletal injury (MSKI) risk is increased following RTD/A after concussion. However, despite the well-documented increased MSKI risk following concussion, the underlying neuromuscular mechanisms contributing to this increased risk have yet to be definitively determined. The underlying mechanism contributing to increased MSKI risk is likely a multifaceted issue that requires a comprehensive study to identify all of the factors.

Understanding the neuromuscular control deficits that persist after concussion and how these deficits change over time (longitudinally) will greatly expand the existing knowledge of why individuals are at greater MSKI risk following concussion. Thus, the overall objective is to elucidate the neuromuscular control mechanisms that contribute to increase MSKI risk following concussion so that effective MSKI risk mitigation strategies can be developed. The study team hypothesizes that concussed individuals will display aberrant neuromuscular control function that increases MSKI risk, as compared to non-concussed controls.

This study will address the following specific aims:

Specific Aim #1: Determine the neuromuscular control factors that differ between concussed and non-concussed military Service Members and physically active civilians that may contribute to MSKI risk after concussion.

Hypothesis #1: Concussed individuals will display aberrant neuromuscular functioning (e.g., atypical joint loading, slower time to stabilization, lower muscular twitch interpolation) that increases MSKI risk after reporting asymptomatic as compared to non-concussed controls.

Specific Aim #2: Determine the differences in patient reported outcome (PRO) measures between military Service Members and physically active civilians with and without concussion.

Hypothesis #2: Concussed individuals will report worse functioning on PRO measures (e.g., National Institutes of Health Patient-Reported Outcomes Measurement Information System [PROMIS] and psychological resiliency) as compared to non-concussed matched controls.

Exploratory Aim #1: Determine the time-dependent changes in neuromuscular control factors following concussion (initial, 6-week post-initial, 12-week post-initial) for concussed and non-concussed military Service Members and physically active civilians.

Exploratory Hypothesis #1: Concussed individuals will display greater changes, regressing toward the non-concussed population, in neuromuscular control (e.g., joint loading, time to stabilization, muscular twitch interpolation) from initial-to-6-week and initial-to-12-week measures as compared to non-concussed controls (anticipate non-significant changes).

This is a multi-center prospective, case-matched control observational study to identify the differences in neuromuscular function following concussion that may contribute to increased MSKI risk. A convenience sample of concussed Service Members and physically active civilians who self-report being asymptomatic and gender, age, occupation, and physical activity matched non-concussed controls will complete the study procedures described below: 1) within 5 days of being asymptomatic ("initial"); 2) 6 weeks post-initial neuromuscular control assessment ("6-week post-initial"; ±72 hours); and 3) 12 weeks post-initial neuromuscular control assessment ("12-week post-initial"; ±72 hours).

Concussed and non-concussed matched control participants will complete the same dynamic movement assessment, neuromuscular testing, and sensory assessment batteries. Control participants will complete the battery at the same time intervals as their concussed counterpart, ± 72 hours. Full-body kinematics will be tracked via stereophotogrammetric motion capture systems and kinetic measures will be captured via 6-degree-of-freedom force platforms. Peak isometric strength and voluntary muscle activation, via the interpolated twitch technique (ITT), and muscular ramp contraction assessment of the dominant and non-dominant knee extensors and plantar flexors will be assessed via a dynamometer (WRNMMC: Baltimore Therapeutic Equipment (BTE) Primus RS [Baltimore Therapeutic Equipment, Maryland and Colorado, USA]; UGA: Biodex System 4 [Biodex Medical Systems, Shirley, New York, USA]). The sensory assessments will examine proprioception (sensation of joint movement) and light touch sensation. The proprioception assessments will utilize the three-dimensional motion capture equipment (closed chain) and the dynamometer (passive joint repositioning). The light touch sensation will utilize Semmes-Weinstein Monofilaments to assess the participant's ability to detect various sensory thresholds on the foot. Additionally, study participants will self-report any MSKI they sustain and psychosocial measures monthly for up to 1-year following the initial neuromuscular control assessment.

Data and Statistical Analysis Plan

Data will be collapsed across trials for all for multi-trial assessments for each data collection time point (initial, 6-Week post-initial, 12-Week post-initial). The time from initial concussion diagnosis until the first data collection time point ("initial"), over-ground gait velocity, and potentially limb dominance will be utilized as a covariates for all statistical analyses. Other covariates, including gender, age, occupation, and physical activity will be explicitly controlled between groups by the matching procedure used in the study design and will therefore be unlikely to contribute to any observed effects; however, the study team will evaluate the importance of these variables in each analysis. These covariates will initially be included in each model, when appropriate; however, if a covariate accounts for little or no variance (p > 0.2), it will be removed from the models. For all statistical analyses, statistical significance will be set a priori as α ≤ 0.05.

For Specific Aim #1, generalized linear mixed effects models including the fixed effects of study group (concussed group; non-concussed control group) and the random (subject-level) effect of participant will determine whether there is a statistically significant difference between concussed and non-concussed matched controls in each biomechanical outcome collected during the movement assessments, while accounting for the aforementioned covariates. Models will be generated for each movement assessment. Additionally, the models exploring gait variables will include task complexity (single-task vs dual-task) to determine whether there is a statistically significant difference in performance in regards to task complexity.

For Specific Aim #2, generalized linear models including group (concussed group; non-concussed control group) as the independent variable and each PRO as the dependent variable to determine whether there is a statistically significant difference in self-reported function and symptoms between concussed and non-concussed matched controls for each PRO. These models will include similar covariates as were used to analyze Specific Aim #1. For ordinal outcomes, the study team will use cumulative link models.

For Exploratory Aim #1, generalized linear mixed effects models treating time as both a fixed effect and including a random slope of time by participant, and fixed effects of group (concussed and non-concussed matched control), time point (initial, 6-Week post-initial, 12-Week post-initial), the interaction of group and time, as well as other covariates as previously described will determine whether there is a statistically significant difference between concussed and non-concussed matched controls in the outcomes of interest over time. Planned comparisons will evaluate between group differences at each time point. The study team will also analyze loss to follow up ("attrition"), to identify if any trends in performance on any of the biomechanical measures or PRO relate to the likelihood of study dropout. If no trends in missing data are observed, participants with at least one follow-up session will be included in all analyses.

ELIGIBILITY:
Inclusion Criteria:

Concussed Cohort

* 18-40 years old.
* Self-reported asymptomatic post-concussion following enrollment into the study and monitoring of symptoms by research personnel via daily self-reported symptom questionnaires.
* Recruited within 5 days following being diagnosed with a concussion, and at least 72 hours prior to self-reporting as asymptomatic.
* Access to a functional email address and the internet for completion of patient reported outcomes (PROs) and musculoskeletal injury measures.

Non-Concussed Cohort

* 18-40 years old.
* Active duty Service members and physically active civilians.
* No self-report history of concussion within the previous 5 years.
* No lingering post-concussion signs/symptoms.
* Same gender as the matched concussed participant.
* Within ±5% of the matched concussed participant's height, weight, and body mass index.
* Within ±2 years of age of the matched concussed participant.
* Participant in the same physical activities (work, recreational sports, average type [no impact, low-impact, high-impact] and duration of physical activity)

Exclusion Criteria:

* Post-Concussion Cohort AND Healthy Non-Concussed Cohort

  * Unable to read or comprehend the English language.
  * Admitted to the hospital following concussion.
  * Sustained a concussion not related to physical activity participation (e.g., blast-related injury, fall from a ladder, motor vehicle accident).
  * Loss of consciousness longer than 30 minutes.
  * Alteration in consciousness longer than 24 hours.
  * Post-traumatic amnesia lasting longer than 1 day.
  * Glasgow Coma Scale below 13.
  * Abnormal brain imaging findings.
  * Sustained a concussion that took longer than 21 days for the individual to report as asymptomatic.
  * A MSKI within the last 6 months that resulted in altered or missed physical activity for 3 or more consecutive days.
  * History of MSKI surgery.
  * Pregnant females (will be eligible for participation in the study once medically cleared to RTD/A by a qualified and licensed healthcare provider following the end of the pregnancy).
  * Participants will be excluded if they present any known contraindications for electrical stimulation. These contraindications include conditions such as: active deep vein thrombosis/thrombophlebitis, any acute injury with concurrent inflammation, hemorrhagic conditions, impaired circulation, impaired local sensations, presence of infection (osteomyelitis, tuberculosis), malignancy, recently radiated tissue, skin disease/damage and/or at-risk skin.
  * Present with any implanted pacemaker, electronic device, or plastic/cement material

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Concussed Cohort: Convenience sample of healthy active duty Service members and physically active civilians who self-report being asymptomatic following a concussion.
  Non-Concussed Cohort: Convenience sample of non-concussed matched active duty Service members and physically active civilians.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Jump-Landing Kinematic and Kinetic Measures | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  The participant will stand on a 30cm tall box, set at a distance that is equal to 50% of the participant's height behind a set of force platforms. Once the participant receives a visual stimulus, he/she will jump so that both feet leave the box at the same time. Upon landing the participant will immediately jump vertically for maximal height. Participants will complete 5 jump-landings. Whole body biomechanics will be collected and kinematic and kinetic measures will be identified at initial ground contact ("initial contact"), the peak angle ("max") during the "landing phase" of the initial landings of the jump-landing, and the difference between these angles ("displacement").
Changes in Single Leg Hop Kinematic and Kinetic Measures | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  The participant will stand on a 30cm tall box, set at a distance that is equal to 50% of the participant's height behind a set of force platforms. Once the participant receives a visual stimulus, he/she will jump so that both feet leave the box at the same time. The participant will jump off the box and land on a single leg with hands on hips. Participants will be instructed to come to a stable position as quickly as possible upon landing. Participants will perform 5 single leg hop trials on each leg (10 total trials). Whole body biomechanics will be collected and kinematic and kinetic measures will be identified at initial ground contact ("initial contact"), the peak angle ("max") during the "landing phase" of the initial landings of the single leg-hop, and the difference between these angles ("displacement").
Changes in Anticipated Cut Kinematic and Kinetic Measures | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  The participant will stand on a 30cm tall box, set at a distance that is equal to 50% of the participant's height behind a set of force platforms. Once the participant receives a visual stimulus, he/she will jump so that both feet leave the box at the same time. The participant will jump off the box and land on a single leg. Immediately upon landing, the participant will cut at a 45° angle (marked with tape on floor) in the direction provided by the study team prior to the trial (cut towards dominant = land on non-dominant foot; cut towards non-dominant = land on dominant foot). Participants will complete 5 trials cutting in each direction (10 total trials). Whole body biomechanics will be collected and kinematic and kinetic measures will be identified at initial ground contact ("initial contact"), the peak angle ("max") during the "landing phase" of the initial landings of the anticipated cutting tasks, and the difference between these angles ("displacement").
Changes in Single-Task Gait Kinematic and Kinetic Measures | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  Participants will complete over-ground gait trials at self-selected walking speed. Participants will start approximately 3m in front of the force platforms so that he/she is at a steady walking speed by the time the participant's foot makes contact with a force platform. No verbal instructions will be provided to indicate that clean foot strikes are required, and participants will be instructed to look straight ahead while walking (i.e., minimizing "targeting"). Participants will complete 5 gait trials so that each foot makes contact with the force platform (10 total trials) for both tasks. Gait velocity, center of mass displacement, and center of mass velocity will be collected from these tasks.
Changes in Dual-Task Gait Kinematic and Kinetic Measures | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  Participants will complete over-ground gait trials as well as gait tasks under a dual-task condition at self-selected walking speed. Participants will start approximately 3m in front of the force platforms so that he/she is at a steady walking speed by the time the participant's foot makes contact with a force platform. No verbal instructions will be provided to indicate that clean foot strikes are required, and participants will be instructed to look straight ahead while walking (i.e., minimizing "targeting"). During dual-task conditions participants will complete Serial Sevens, Serial Nines, etc. Participants will start counting at a randomly generated number between 80 and 120 and will count backwards by the designated denomination. Participants will complete 5 gait trials so that each foot makes contact with the force platform (10 total trials) for both tasks. Gait velocity, center of mass displacement, and center of mass velocity will be collected from these tasks.
Changes in Interpolated Twitch Technique Measurements | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  Participants will be seated in the dynamometer so that the axis of rotation of the participants' dominant knee coincides with the servomotor. Participants will be secured to the chair using seat belts along the chest, waist, and ankle. Adhesive stimulating electrodes will be placed on the skin overlying the distal vastus medialis muscle and proximal vastus lateralis muscle of the thigh on the dominant leg and will be controlled by electrical stimulators. Participants will perform a maximal voluntary isometric contraction (MVIC). During the MVIC, the muscle group will be stimulated with a paired-pulse stimulation, and the increase in torque over the MVIC level (i.e., interpolated twitch torque [ITT]) will be recorded. Following the MVIC, the paired-pulsed stimulation will be administered again (twice) to the relaxed muscle to determine peak electrically-evoked twitch torque (EET).
Changes in Muscular Ramp Contraction Measurements | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  Participants will be seated in the dynamometer so that the axis of rotation of the participants' dominant knee coincides with the servomotor. Participants will be secured to the chair using seat belts along the chest, waist, and ankle. Adhesive stimulating electrodes will be placed on the skin overlying the distal vastus medialis muscle and proximal vastus lateralis muscle of the thigh on the dominant leg, and will be controlled by electrical stimulators. Participants will perform three maximal voluntary isometric contractions (MVIC). The maximal voluntary muscle torque will be determined from this initial test and then used to create a ramping protocol in which the participant will ramp from 20 -100% maximal voluntary contraction over a 2.5 second period.
Changes in Closed-Chain Proprioception | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  The participant will stand with feet shoulder-width apart, feet (toes) pointed anteriorly, heels on the floor, and hands clasped in front of the participants chest. Participants will be asked to squat in a deep, slow, and controlled manner, to what they believe is 60-degrees of knee flexion and to hold that position for 5 seconds. Participants will then return to a full, upright position, march in place 10 times (5 each leg), and regain the original starting position. Participants will then be asked to replicate the same knee joint angle as they did in their initial trials. Participants will perform 3 trials following the initial trial (4 total trials).
Changes in Passive Joint Repositioning | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing,
  Participants will be assessed using the passive motion and direction threshold method on a research dynamometer that passively moves the participant's dominant leg until the minimal detectable change in joint angle is perceived. Participants will be secured to the dynamometer while blindfolded and listening to static noise through headphones to eliminate movement cues. Initial starting positions will be 10° and 125° of knee flexion while the dominant knee will be passively moved at 5°/sec in either flexion or extension directions. The participant will be instructed to hit the "stop" button on the dynamometer once he/she perceives any movement, locking the dynamometer moment arm from moving and while the joint angle is recorded. Participants will perform 2 trials for each range (9 total trials).
Changes in Light Touch Sensation | Initial testing after reporting asymptomatic post-concussion, 6-Weeks post-initial testing, and 12-Weeks post-initial testing.
  Participants will be assessed using Semmes-Weinstein Monofilaments via a "4-2-1" stepping protocol using 20 force-calibrated nylon threads to assess sensory detection thresholds. Participants will lay prone on a treatment table, with their shoe and sock off of their dominant foot, listening to static noise through headphones, while the threads are applied until a "C" shaped bend occurs and is held for 1 second. The threads will be applied using a standard "4-2-1" stepping protocol for one trial. The light touch sensation main outcome measure is the diameter of the thread on the final application.
Changes in Self-Reported Musculoskeletal Injuries | Monthly, through study completion (an average of 1 year)
  Participants will report all of their previous MSKI sustained within 1- year prior to enrollment into the study and any "severe" MSKI they have sustained that resulted in 3 or more consecutive weeks of missed physical activity. Participants will also self-report if they sustain any new MSKIs during the study follow-up period. MSKIs will be operationally defined as: 1) a MSKI that required the participant to seek medical attention from a healthcare provider; or 2) a MSKI that required the participant to not participate in normal physical activity for 3 or more consecutive days. The following information will be self-reported for each injury: 1) date of injury; 2) activity at the time of injury; 3) mechanism of injury (overuse, traumatic); 4) if the injury is recurrent (i.e., previously experienced); and 5) if the MSKI resulted in less than or more than 1 week of missed or altered physical activity.
Changes in NIH-PROMIS Physical Function | Monthly, through study completion (an average of 1 year)
  Physical Function measures an individual's self-reported capabilities rather than his/her actual performance of physical activities. The assessment includes functioning of an individual's upper and lower extremities and neck and spine across a variety of activities.
Changes in NIH-PROMIS Pain Interference | Monthly, through study completion (an average of 1 year)
  Pain Interference measures an individual's self-reported consequences of pain on one's life over the past 7 days. This includes the extent to which pain hinders social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items that assess sleep and enjoyment of life.
Changes in NIH-PROMIS Depression | Monthly, through study completion (an average of 1 year)
  Depression measures an individual's self-reported negative mood, views of self, social cognition, and decreased positive affect and engagement over the past 7 days.
Changes in NIH-PROMIS Anxiety | Monthly, through study completion (an average of 1 year)
  Anxiety measures an individual's self-reported fear, anxiousness, hyperarousal, and somatic symptoms related to arousal (e.g., racing heart) over the past 7 days.
Changes in the Brief Resilience Scale (BRS) | Monthly, through study completion (an average of 1 year)
  A patient's psychological resiliency, their ability to "bounce back or recover from stress" may mediate health outcomes. Psychological resiliency has been associated with patient outcomes following shoulder stabilization surgery within a military population. Individuals who were more resilient had better outcomes (i.e., less time on limited duty status, less attrition from military service) than individuals who were non-resilient. The BRS has moderate test-retest reliability (ICCrange = 0.62-0.69) and has been validated against a number of different scales that measure various aspects of psychological resilience (rrange = -0.68-0.69).
Changes in the Tampa Scale of Kinesiophobia | Monthly, through study completion (an average of 1 year)
  The Tampa Scale of Kinesiophobia (TSK-11) measures pain-related fear of movement and re-injury. Kinesiophobia is an important factor in determining who will successfully RTD/A following a musculoskeletal injury. Kinesiophobia may impact sensorimotor function and movement quality in dynamic environments, potentially increasing musculoskeletal injury risk.

CONTACTS AND LOCATIONS:
Overall Officials: Bradford D Hendershot, PhD, Principal Investigator — Walter Reed National Military Medical Center; Robert C Lynall, PhD, Study Director — University of Georgia; Timothy C Mauntel, PhD, Study Director — Womack Army Medical Center
Locations (3):
- United States (3):
  - University of Georgia, Athens, Georgia
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lynall RC, Wasser JG, Brooks DI, Call JA, Hendershot BD, Kardouni JR, Schmidt JD, Mauntel TC. Investigating post-mild traumatic brain injury neuromuscular function and musculoskeletal injury risk: A protocol for a prospective, observational, case-controlled study in service members and active individuals. BMJ Open. 2023 Mar 22;13(3):e069404. doi: 10.1136/bmjopen-2022-069404. PMID 36948547

DOCUMENTS (1):
  • Informed Consent Form (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT05122728/ICF_000.pdf